CLINICAL TRIAL: NCT01204099
Title: Phase 1/2 Study of PX-866 and Docetaxel in Patients With Solid Tumors
Brief Title: Study of PX-866 and Docetaxel in Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cascadian Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PX-866-002
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2015-04

CONDITIONS: Non Small Cell Lung Cancer (NSCLC); Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Keywords: PX-866; Non small cell lung cancer; solid tumors; Squamous cell cancer of the head and neck; docetaxel; NSCLC; taxotere; SCCHN; PI-3K; PI3 kinase; PI3K
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Hereditary Sensory and Autonomic Neuropathies | interventions — Docetaxel; PX-866

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Docetaxel (NSCLC) (Active Comparator): IV docetaxel administered once every three weeks as per standard of care. Treatment continues until disease progression, unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: Docetaxel
- PX-866 (NSCLC) (Experimental): Oral PX-866 administered daily at the RD in combination with IV docetaxel administered once every three weeks on a 21 day cycle. Treatment continues until disease progression, unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: Docetaxel; Drug: PX-866
- Docetaxel (SCCHN) (Active Comparator): IV docetaxel administered once every three weeks as per standard of care. Treatment continues until disease progression, unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: Docetaxel
- PX-866 (SCCHN) (Experimental): Oral PX-866, administered daily at the RD in combination with IV docetaxel administered once every three weeks on a 21 day cycle. Treatment continues until disease progression, unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: Docetaxel; Drug: PX-866

INTERVENTIONS:
Drug: Docetaxel
  Other Names: taxotere
Drug: PX-866
  Arms: PX-866 (NSCLC); PX-866 (SCCHN)

SUMMARY:
Phase 1: To determine the maximally tolerated dose (MTD) or recommended dose (RD) and any potential efficacy of PX-866 in combination with docetaxel in patients with solid tumors.

Phase 2: To determine the antitumor activity and safety of PX-866 in combination with docetaxel versus docetaxel alone in patients with NSCLC or SCCHN.

DETAILED DESCRIPTION:
This is a Phase 1/2 open-label study. In the Phase 1 part of the study, PX-866 was given in combination with docetaxel to patients with incurable locally advanced, recurrent or metastatic cancer.

Phase 2 of the study is an open-label, randomized evaluation of the antitumor activity and safety of PX-866, administered at the MTD/RD identified in Phase 1 (8mg daily), in combination with docetaxel versus docetaxel alone in patients with locally advanced, recurrent, or metastatic NSCLC (Group 1) or patients with locally advanced, recurrent, or metastatic SCCHN (Group 2).

Group 1 (patients with locally advanced, recurrent, or metastatic NSCLC) is now closed to enrollment.

All treatments will be administered on a 21-day cycle. Docetaxel 75 mg/m2 will be administered IV on Day 1 of each 21-day cycle. PX-866 will be administered orally or via PEG tube (if applicable) once per day on Days 1 to 21 of all treatment cycles in patients randomized to the treatment arm containing PX-866.

Patients will be evaluated for progression approximately every 6 weeks. Patients with stable disease (SD) or better, per investigator assessment, will receive repeat cycles of treatment on a 21-day schedule until disease progression, unacceptable toxicity or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years at time of consent
* Agrees to use a medically accepted form of contraception from the time of consent to completion of all follow up study visits
* If female of child bearing potential, negative pregnancy test (not required for post menopausal females)
* Signed an informed consent document that has been approved by an institutional review board or independent ethics committee (IRB/IEC)
* Has either locally advanced, recurrent, or metastatic NSCLC for which they have received at least 1 and no more than 2 prior systemic treatment regimens that may include up to 1 platinum based chemotherapy regimen and/or an epidermal growth factor receptor (EGFR) inhibitor OR locally advanced, recurrent or metastatic SCCHN for which they have received at least one and no more than two prior systemic treatment regimens.
* Measurable disease per Response Evaluation Criteria In Solid Tumors
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* In the opinion of the clinical investigator, life expectancy >3 months
* Adequate hematologic function as defined by:

  * Hemoglobin ≥ 9 g/dL
  * Absolute neutrophil count (ANC) ≥1500 cells/µL
  * Platelets ≥100,000/µL
* Adequate hepatic function as defined by the following:

  * Bilirubin ≤ ULN
  * Aspartate aminotransaminase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤1.5 x upper limit of normal (ULN)
* Creatinine level ≤1.5 x ULN

Exclusion Criteria:

* Has medical, social, or psychosocial factors that, in the opinion of the investigator, could impact safety or compliance with study procedures
* Is breastfeeding
* Treatment with any systemic chemotherapy, epidermal growth factor receptor (EGFR) inhibitor, radiation or experimental agent within 4 weeks of study drug dosing. Washout period following palliative radiation should be discussed with the study medical monitor
* Previous treatment with docetaxel except for patients in Phase 2 who received a docetaxel containing regimen as part of adjuvant or neoadjuvant therapy which was completed at least 6 months prior to study drug dosing
* Previous treatment with a phosphatidylinositol 3 kinase (PI 3K) inhibitor
* Known human immunodeficiency virus (HIV)
* Known or suspected clinically active brain metastases. Previously treated and stable brain metastases are allowable. Stable brain metastases are defined as no change on CT scan or MRI for minimum of two months AND no change in steroid dose for a minimum of four weeks, unless change due to intercurrent infection or other acute event
* Grade >2 peripheral neuropathy, as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.02
* Any other significant medical or psychiatric condition that in the opinion of the investigator renders the patient inadequate for participation
* History of severe hypersensitivity reactions to docetaxel or to other drugs formulated with polysorbate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 42 days

SECONDARY OUTCOMES:
Objective response rate (ORR) | 42 days
Incidence and severity of adverse events | 42 days
Overall survival | 42 days

CONTACTS AND LOCATIONS:
Locations (33):
- United States (29):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Southwest Cancer Care, Escondido, California
  - Bay Area Cancer Research Group, LLC, Pleasant Hill, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Eastern Colorado Health Care System - Denver VA, Denver, Colorado
  - Cancer Center of Pasco-Pinellas, Holiday, Florida
  - Cancer Center of Kansas, Wichita, Kansas
  - John Hopkins University, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Oncology, Hematology, Latham, New York
  - Beth Israel Hospital, New York, New York
  - New York University Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Northwest Cancer Specialists, Tualatin, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Oncology - South Austin, Austin, Texas
  - Mary Crowley Cancer Center, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Oncology and Hematology Associates of SW Virginia, DBA Blue Ridge Cancer Care, Christiansburg, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Columbia Basin Hematology & Oncology, Kennewick, Washington
  - Medical Oncology Associates, Spokane, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
- Canada (4):
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - London Regional Cancer Program, London, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - CHUS Hopital Fleurimont, Sherbrooke, Quebec